CLINICAL TRIAL: NCT07088549
Title: Effect of Continuous Interstitial Glucose Monitoring on Glycaemic Targets and Clinical Outcomes in Critically Ill
Brief Title: Intermittent Versus Continuous Glucose Monitoring in Intensive Care Unit
Acronym: ICONS-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Peter Radsel, Head of Clinical Department of Internal Intensive Care Medicine, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ICONS-ICU
Record Dates: First submitted 2025-06-23; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness; Hyperglycaemia; Hypoglycaemia
Keywords: continuous glucose monitoring; icu
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CGM monitoring (Active Comparator): DexcomG7 continuous glucose monitor
  Interventions: Device: Continuous glucose monitoring
- Standard of care (Active Comparator): Radiometer ABL800 blood glucose measurement
  Interventions: Diagnostic Test: Control Arm - standard of care

INTERVENTIONS:
Device: Continuous glucose monitoring — Intravenous insulin therapy will be guided by interstitial glucose measurements using DexcomG7 continuous glucose monitor. Confirmatory blood glucose tests will be performed daily. In extreme clinical conditions (post-resuscitation, pH < 7.20, severe hypoxia, severe haemodynamic compromise), confirmatory blood tests will be performed in 2 hour intervals until clinical improvement.
  Arms: CGM monitoring
Diagnostic Test: Control Arm - standard of care — Intravenous insulin dosing will be guided according to blood glucose measurements using RadiometerABL800 (standard of care). DexcomG7 continuous glucose monitor will be applied in blinded mode for interstitial glucose monitoring for later CGM metrics and comparison analysis.
  Arms: Standard of care

SUMMARY:
Glucose control is an important part of supportive care for critically ill patients. Achieving optimal glucose control in such situations is challenging due to frequent fluctuations in blood glucose levels. These changes are often difficult to detect because the monitoring procedures are complex and require significant staff involvement, frequent blood draws, and consequent blood loss. Continuous glucose monitoring (CGM) is a simple and minimally invasive technique that has been approved and increasingly used by people with diabetes mellitus. However, its effectiveness in terms of glucose control management and accuracy in conditions with severe organ dysfunction has not been established.

The goal of this study is to assess the performance of CGM-guided glucose control in comparison to the standard glucose monitoring procedure. Additionally, the accuracy of CGM measurements under critical conditions will be evaluated against the standard of care.

DETAILED DESCRIPTION:
This study will be an investigator-initiated, non-commercial, prospective, single-center, parallel-group, randomized controlled trial. Critically ill patients with hyperglycemia requiring intravenous insulin therapy will be randomly assigned to two groups: an intervention group that will receive intravenous insulin therapy aided by continuous glucose monitoring (CGM) measurements and a control group that will receive intravenous insulin therapy guided by arterial blood glucose measurements (RadiometerABL800). Patients will be enrolled within 48 hours after ICU admission. Intravenous insulin dosing will be adjusted according to the in-house glycaemic management protocol. After enrollment, patients will be monitored for maximal 10 days (duration of the sensor) or until stopping intravenous insulin therapy, ICU discharge or death, whichever occurs first, if these events happen before the sensor duration ends.

The primary outcome of the study will be the proportion of time spent within the target range of 7.8-10.0 mmol/L. Secondary outcomes will include mean glucose levels and other CGM metrics, daily vasoactive-inotropic score calculation, hospital length of stay, hospital-acquired infections, and acute renal failure.

Additionally, an accuracy analysis in extreme clinical conditions (pH < 7.20, post-resuscitation, ECMO support, severe haemodynamic instability, hypoxia) will be performed by comparing CGM measurements measured by DexcomG7 with arterial blood glucose measurements (RadiometerABL800) from the electronic health record. Satisfaction of health-care personnel will be evaluated. Sensor-related complications will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* admission to the level 3 ICU
* two consecutive blood glucose measurements > 10.0 mmol/L
* intravenous insulin therapy

Exclusion Criteria:

* expected ICU stay < 48 hours
* pregnancy
* type 1 diabetes
* diabetic emergencies (DKA, DAHS)
* severe skin disease
* severe neutropenia (< 0.5 × 10^9/L)
* severe coagulopathy (thrombocytes < 20 × 10^9/L)
* manufacturer-defined conditions (hydroxyurea use, acetaminophen more than 4 g daily)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time in range 7,8 - 10,0 mmol/l | from the enrollment until completion of the continuous glucose monitoring (up to 10 days)
  Percentage of time within recommended glucose range

SECONDARY OUTCOMES:
Mean glucose levels | from the enrollment until completion of the continuous glucose monitoring (up to 10 days)
Glycemic variability | from the enrollment until completion of the continuous glucose monitoring (up to 10 days)
  assessed by the coefficient of variation (CV) and standard glucose variation
Vasopressor inotropic score | from the enrollment until completion of the continuous glucose monitoring (up to 10 days)
  estimated amount of vasopressor support, daily calculated with the Vasoactive Inotropic Score (VIS): minimum 0 - 5 points (low doses), maximum > 45 points (highest doses)
Hospital acquired infections | from the enrollment until hospital discharge, approximately 30 days
  pneumonia, bloodstream infections, urinary infections
Acute renal failure | from the enrollment until hospital discharge, approximately 30 days
  defined by AKIN (acute kidney injury) classification

OTHER OUTCOMES:
Hospital mortality | from the enrollment and before hospital discharge, approximately 30 days
  death during hospitalization
Time above range (level 1 and 2) | from the enrollment until completion of the continuous glucose monitoring (up to 10 days)
  percentage of time above 10,1 - 13,9 mmol/l (level 1) and above 13,9 mmol/l (level 2)
Time below range (level 1 and 2) | from the enrollment until completion of the continuous glucose monitoring (up to 10 days)
  percentage of time below 3,0 - 3,8 mmol/l (level 1) and below 3,0 mmol/l (level 2)

CONTACTS AND LOCATIONS:
Overall Officials: Milica Lukic, MD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: 1 month after publication End date: no end date
Access Criteria: IPD and supporting information will be stored and shared in the Repository of the University of Ljubljana, Slovenia. Access will be provided on request by the Repository.